CLINICAL TRIAL: NCT04644770
Title: A Phase 1 Study of JNJ-69086420, an Actinium-225-Labeled Antibody Targeting Human Kallikrein-2 (hK2) for Advanced Prostate Cancer
Brief Title: A Study of JNJ-69086420, an Actinium-225-Labeled Antibody Targeting Human Kallikrein-2 (hK2) for Advanced Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108817; 69086420PCR1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms; Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation (Experimental): Participants will receive JNJ-69086420 with one or multiple doses. The dose levels will be escalated based on the dose limiting toxicities (DLT) evaluation by Study Evaluation Team (SET) until the recommended Phase 2 Dose (RP2D) has been identified.
  Interventions: Drug: JNJ-69086420
- Part 2: Dose Expansion (Experimental): Participants in one or more cohorts will receive JNJ-69086420 at the RP2D(s) determined in Part 1.
  Interventions: Drug: JNJ-69086420
- Part 3: Combination Therapy (Experimental): Participants will receive JNJ-69086420 at the determined RP2D(s) and fixed dose of JNJ-78278343.
  Interventions: Drug: JNJ-69086420; Drug: JNJ-78278343
- Part 4: HSPC Expansion (Experimental): Participants with HSPC will receive JNJ-69086420 at the RP2D(s) in Part 4(a), and JNJ-69086420 following stereotactic body radiation therapy in Part 4(b).
  Interventions: Drug: JNJ-69086420; Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Drug: JNJ-69086420 — Participants will receive JNJ-69086420.
  Other Names: Actinium-225-DOTA-h11B6
Drug: JNJ-78278343 — Participants will receive JNJ-78278343.
  Arms: Part 3: Combination Therapy
Radiation: Stereotactic body radiation therapy — Participants will receive stereotactic body radiaition therapy.
  Arms: Part 4: HSPC Expansion

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose(s) (RP2D[s]) of JNJ-69086420 in Part 1 (Dose Escalation), to determine safety and preliminary signs of clinical activity at the RP2D(s) in Part 2 (Dose Expansion), to determine safety of JNJ-69086420 at the RP2D(s) as a combination therapy in Part 3 (combination therapy) and to determine safety of JNJ-69086420 at the RP2D(s) in participants with metastatic hormone-sensitive prostate cancer (mHSPC) in Part 4.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1, Part 2, Part 3: Metastatic castration resistant prostate cancer (mCRPC) with histologic confirmation of adenocarcinoma (adenocarcinoma with small-cell or neuroendocrine features is allowed) with prior exposure to at least one androgen receptor (AR) targeted therapy (for example [e.g.], abiraterone acetate, enzalutamide, apalutamide, darolutamide). In addition: Part 1: prior taxane or other chemotherapy is acceptable but not required. Part 2a: prior taxane or other chemotherapy required, Part 2b: no prior taxane or other chemotherapy, Part 2c: mCRPC that has progressed after prior treatment with lutetium Lu-177 vipivotide tetraxetan, with or without prior chemotherapy, Part 3: prior taxane or other chemotherapy is acceptable but not required & For Part 4a: metastatic HSPC, For Part 4b: disease that can be treated with less than or equal to (<=) 5 radiation fields and no visceral metastases
* Parts 1, 2 & 3: Prior orchiectomy or medical castration, or, for participants who have not undergone orchiectomy, must be receiving ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analog (agonist or antagonist) prior to the first dose of study drug and must continue this therapy throughout the treatment phase. This criterion does not apply to Part 4
* Palliative radiotherapy (e.g. soft tissue lesions) must be completed greater than (>) 2 weeks prior to start of study drug except for palliative radiotherapy for pain (e.g., bone pain), which may be used any time prior to first dose
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ functions as reflected in laboratory parameters

Exclusion Criteria:

* Prior treatment with radium Xofigo (Ra 223 dichloride), strontium, samarium, or other radioconjugate therapy, other systemic anti-neoplastic therapy <=30 days prior to the first dose of study drug except for luteinizing hormone-releasing hormone agonists/antagonists or GnRH agonists/antagonists. Novel androgen axis drugs <=14 days prior to the first dose of study drug. In addition: Part 2b: Must not have received prior treatment with chemotherapy (eg, docetaxel) or poly ADP ribose polymerase (PARP) inhibitors, Part 2c: Prior treatment with lutetium Lu-177 vipivotide tetraxetan is required, but must have been completed >42 days prior to first dose of study drug, Part 3: Must not have received prior treatment with JNJ-78278343, Part 4: Must not have received ADT or AR-targeted therapy less than or equal to (<=) 56 days prior to first dose of study drug
* Known history of myelodysplastic syndrome, leukemia, or hematological malignancy with features suggestive of myelodysplastic syndrome/acute myeloid leukemia at any timepoint
* Toxicity from prior anticancer therapy has not resolved to baseline levels or to Grade <= 1 (except alopecia, radiation tissue fibrosis, or peripheral neuropathy)
* Known allergies, hypersensitivity, or intolerance to JNJ-69086420 or its excipients and protein therapeutics. For Part 3, known allergies, hypersensitivity, or intolerance to JNJ-78278343 or its excipients or protein therapeutics
* Active or chronic hepatitis B or hepatitis C infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 2 years and 4 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | Up to 2 years and 4 months
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Number of Participants with AEs by Severity | Up to 2 years and 4 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.

SECONDARY OUTCOMES:
Percentage of Participants with Prostate Specific Antigen (PSA) Response | Up to 2 years and 4 months
  PSA response rate is defined as the percentage of participants with a decline of PSA of 50 percent (%) or more from baseline and that is subsequently confirmed.
Overall Response Rate (ORR) | Up to 2 years and 4 months
  ORR is defined as the percentage of participants who have a Partial Response (PR) or better according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 without evidence of bone progression according to Prostate Cancer Working Group 3 (PCWG3).
Maximum Observed Serum Concentration/Radioactivity (Cmax) of JNJ-69086420 | Up to 2 years and 4 months
  Cmax is defined as the maximum observed serum concentration/radioactivity of JNJ-69086420.
Time to Reach Maximum Observed Serum Concentration/Radioactivity (Tmax) of JNJ-69086420 | Up to 2 years and 4 months
  Tmax is defined as time to reach maximum observed serum concentration/radioactivity of JNJ-69086420.
Area Under the Serum Concentration-time Curve From Time Zero to t Time (AUC[0-t]) of JNJ-69086420 | Up to 2 years and 4 months
  AUC(0-t) is defined as the area under the serum concentration-time curve from time zero to t of JNJ-69086420.
Number of Participants With Anti-JNJ-69086420 Antibodies | Up to 2 years and 4 months
  Number of participants with anti-JNJ-69086420 antibodies will be assessed to evaluate the potential immunogenicity.
Part 3: Serum Concentration of JNJ-78278343 | Up to 2 years and 4 months
  Venous blood samples will be collected for assessment of serum concentrations of JNJ-78278343.
Part 3:Number of Participants With Anti-JNJ-78278343 Antibodies | Up to 2 years and 4 months
  Number of participants with anti-JNJ-78278343 antibodies will be assessed to evaluate the potential immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- United States (11):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - East Jefferson General Hospital, Metairie, Louisiana
  - Tulane University Hospital & Clinics, New Orleans, Louisiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Lehner F, Salemi S, Millan C, Kundig C, Eberli D. Inhibition of Growth and Induction of Apoptosis of Human Prostate Cancer Cells by Enzymatic Blockage of Kallikreins. Prostate Cancer. 2026 Jan 11;2026:7871208. doi: 10.1155/proc/7871208. eCollection 2026. PMID 41531507